CLINICAL TRIAL: NCT00338910
Title: Pharmacokinetic Interaction Study Between Budesonide and Metronidazole in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Dr. Falk Pharma GmbH (Industry); Principal Investigator: Univ. Hosp. Tuebingen, Dept. of Clinical Pharmacology (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUC-58/BIO
Record Dates: First submitted 2006-06-19; First posted 2006-06-20 (Estimated); Last update posted 2007-12-11 (Estimated); Status verified 2007-12

CONDITIONS: Healthy
Keywords: healthy volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Budesonide 2 single doses, Metronidazole multiple-dose — Budesonide 3 mg single oral dose on Day 1 and Day 9. Metronidazole 750 mg b.i.d. from Day 2 until Day 8, Metronidazole 750 mg once daily (in the morning) on Day 9.

SUMMARY:
The primary objective of this study is to describe a possible effect of metronidazole on PK of budesonide in healthy volunteers.

DETAILED DESCRIPTION:
The primary objective of this study is to describe a possible effect of metronidazole on PK of budesonide in healthy volunteers.

Secondary objectives:

1. Effect of budesonide on metronidazole steady-state PK (primarily described as area under the concentration-time-curve).
2. Urinary 6β-hydroxycortisol (being a marker of CYP3A activity) and cortisol excretion before and during metronidazole multiple-dose co-administration.
3. Safety parameters.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* Caucasian origin
* Age: between 18 and 55 years (inclusive)
* Body mass index (BMI) within 18-30 kg/m²
* Body weight at least 50 kg, at most 100 kg
* Non-smoker (or ex-smoker ≥1 year), proven by urine cotinine <500 ng/ml
* Clinically acceptable supine blood pressure and pulse rate, i.e. BP 100-145 mmHg systolic, 60-90 mmHg diastolic and pulse rate 50-100 bpm
* Normal ECG
* Participants must perform an adequate contraception during the study and until 6 months after the last dose of the present trial
* Ability to communicate well with the investigator and comply with the requirements of the entire study
* Written consent

Exclusion Criteria:

* Subjects with contraindications for budesonide
* Subjects with contraindications for metronidazole
* History or current clinical evidence of any cardiac, cardio-vascular, pulmonary, gastrointestinal, (cholangio-)hepatic, renal, endocrine, neurological, musculoskeletal, ophthalmological, infectious, haematological, oncological, psychiatric, or other acute or chronic diseases and/or pathological findings which might interfere with the drugs' safety, tolerability, absorption and/or pharmacokinetics
* History or current evidence of clinically relevant allergies or idiosyncrasy to drugs or food
* Clinically relevant abnormalities in clinical chemical, hematological or any other laboratory variables
* Current smoker or ex-smoker ≤ 1 year
* Excessive alcohol consumption (³ 35 g/day in males)
* Abuse of drugs
* Positive drug screening
* Positive anti-HIV-test, HBsAg-test or anti-HCV-test
* Proneness to orthostatic dysregulation, faintings, or blackouts
* Heavy tea or coffee drinkers (more than 1 l ≈ 6 cups per day)
* Administration of glucocorticosteroids within 6 weeks prior to study day 1 or during the trial
* Repeated use of drugs during the last 4 weeks prior to study day 1 or during the trial, which might influence hepatic biotransformation
* Any medication including OTC medication within the last 14 days prior to study day 1 or during the trial (single intake of a drug may be accepted if judged by the investigators to have no clinical relevance and no relevance for the study objectives)
* Intake of grapefruit-containing food or beverages within 7 days prior to study day 1 or during the trial
* Clinically relevant acute or chronic bacterial, fungal or viral infections
* Surgery of the gastrointestinal tract which may interfere with drug absorption (not applicable for minor abdominal surgery such as e.g. appendectomy and herniotomy)
* Vegetarian diet or other peculiar dietary habits which would preclude the subject's acceptance of standardized (non-vegetarian) meals
* Subjects suspected or known not to follow instructions
* Subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to as a result of their participation in the study
* Patients known to be in financial difficulties, which could interfere with their appraisal of the informative instructions
* Vulnerable subjects (e.g., persons kept in detention or persons who are depending on the sponsor or the investigator)
* Blood donation or other blood loss of more than 400 ml within the last 2 months prior to study day 1
* Participation in a clinical trial within the last 2 months prior to study day 1 (assessed by anamnestic inquiry)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-05; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
AUC

SECONDARY OUTCOMES:
other PK parameters

CONTACTS AND LOCATIONS:
Overall Officials: Christoph H Gleiter, MD, Principal Investigator — Department of Clinical Pharmacology